CLINICAL TRIAL: NCT03254316
Title: Healthcare Associated Infection Surveillance in NICU of Assiut University Children's Hospital
Brief Title: Health Care Associated Infection Surveillance in NICU
Status: Completed | Type: Observational
Sponsor: Gehad Salah El-Den Mahmoud Mohammad (Other)
Responsible Party: Sponsor-Investigator, Gehad Salah El-Den Mahmoud Mohammad, Resident doctor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: HCAISN
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Health Care Associated Infection
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Healthcare - Associated Infection Surveillance In Neonatal Intensive Care Unit of Assiut University Children's Hospital.The objective of study is to determine the incidence, infection sites, causative organisms and risk factors related to healthcare-associated infections in NICU in Assiut University Children hospital.

DETAILED DESCRIPTION:
Nosocomial infections (NIs) are a major public health problem worldwide . Nosocomial infections are those acquired in or associated with hospitals. They are also known as hospital-acquired or healthcare-associated infections. The usual deﬁnition of a hospital-acquired infection is one that was not present or incubating when the patient was admitted to a hospital or healthcare facility; where there is doubt, a cut-off period of 48 hours after admission is used.The terms hospital-acquired and healthcare-associated are often used interchangeably, but 'healthcare-associated' also has the wider meaning of any infection acquired as a result of healthcare in any setting.

Nosocomial infections are common, and may be serious or fatal. Some are unavoidable but doctors' duty of care to their patients extends to fundamental matters such as basic hygiene, which may prevent patients becoming infected, and avoidance of unnecessary antibiotics, to discourage development of resistance Health care-associated infections (HC-AIs) are a major cause of morbidity and mortality in neonatal intensive care units (NICUs) and lead to increases in hospital length of stay and treatment cost. Higher nosocomial infection incidence in NICUs was related to longer duration of hospital stay, and invasive interventions and medical treatments. HC-AIs, especially device-associated health care-associated infections (DA-HAIs), were also common in newborns because of their insufﬁcient immune system and mechanical barriers, as well as lack of protective ﬂora

ELIGIBILITY:
Inclusion Criteria:

1. Age at admission ( 0-28 DAY )
2. Neonates who admitted for more than 48 hours

Exclusion Criteria:

1. Age:more than 28days
2. Neonates who admitted for less than 48 hours.
3. Neonates who admitted for infection reasons as (pneumonia, MAS, AGE and skin infection).
4. Neonates with potentially infection (PROM, chorioamnionitis, TOF)
5. Neonates with congenital infections

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a prospective clinical study covered a period of 12 months in a tertiary neonatal intensive care unit in NICU of Assiut university children's hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Detect incidence of nosocomial infection in NICU | 1 year
  To detect impact of nosocomial infection on outcome of neonates admitted in NICU

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Shorat, Professor, Study Director — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Egypt